CLINICAL TRIAL: NCT06491693
Title: Can Ultrasonographic Screening of Optic Sheath Diameter Be an Early Detector of Norological Morbidities Related Carotis Endarterectomy
Brief Title: Can Optic Nerve Sheath Diameter Detect Norological Morbidities for Patients Undergoing Carotis Endarterectomy
Status: Recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Zülfiye Yıldız, principal investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: KAEK-11/22.05.2024.02
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Optic Nerve Sheath Diameter Measurements for Carotis Endarterectomy
Keywords: optic nerve sheath dimater; carotis endarterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main purpose of this study is to investigate the contribution of changes in Optic Nerve Sheath Diameter (OSNC) measured at different periods during Carotid Endarterectomy (CEA) operations to the prediction of neurological problems detected in the postoperative period. The secondary aim of the study is to examine the relationship between optic nerve sheath diameter measurement and other routinely used perioperative follow-up parameters in terms of predicting neurological problems.

DETAILED DESCRIPTION:
CEA operations are generally performed on elderly patients and patients with different comorbidities. These patients have carotid artery stenosis and often thrombus. 85% of all stroke cases are due to ischemic causes, and 15-30% of them are due to carotid artery stenosis. The treatment method is usually surgery. CEA operations. Early detection of cerebral hypoperfusion and ischemia during the operation is important. Carotid clamp applications, which must be used during the operation upon the decision of the surgical team, may cause cerebral hypoperfusion. In addition, the resulting systemic hypotension further worsens this situation. In order to prevent cerebral hypoperfusion, carotid shunt applications can be performed to ensure flow continuity, and at the same time, cerebral hypoperfusion is tried to be prevented by keeping the mean arterial pressure high. Close monitoring of these cases and follow-up of cerebral perfusion adequacy is important to detect ischemia and embolism events that may develop especially during these periods. ECG, blood pressure, oxygen saturation, near infrared spectroscopy (NIRS), and Bispectral index (BIS) are routinely used in monitoring. In addition, it is reported in the literature that there are changes in ONCH, which can be easily evaluated with USG, in cases such as ischemic stroke and increased intracranial pressure, an increasing trend occurs and shows an excellent correlation with invasive intracranial pressure monitoring. ONSD has been associated with increases in intracranial pressure. In these patients in whom a carotid clamp is placed, an increase in intracranial pressure due to ischemia and cerebral hypoperfusion and a corresponding increase in ONSD may be observed. In this context, in our study, in addition to routine monitoring methods, we measured the Optic Nerve Sheath Diameter (OSCN), which can be examined practically with the help of ultrasonography (USG), which we use in our daily practice in the operating room, and does not require any additional cost and labor, and thus, we measured the parameters such as cerebral ischemia and increased intracranial pressure that may develop in the intraoperative period. We planned to investigate its contribution to the prediction of neurological problems and its relationship with other follow-up parameters. Measurement of ONSC with USG is a very simple, noninvasive and non-harmful method.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 50 and 80, who are planned for elective CEA under general anesthesia, who come in a spontaneously breathing, conscious and cooperative state.

Exclusion Criteria:

* Patients who are under 50 years of age, over 80 years of age, have neurological findings caused by reasons other than carotid lesion, and are intubated.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It was planned to include 40 patients, male and female, between the ages of 50 and 80, who were scheduled for elective CEA under general anesthesia, taking into account previous similar studies (1,3,4) and power analysis.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The aim is to investigate the contribution of changes in Optic Nerve Sheath Diameter (OSNC) measured at different periods during Carotid Endarterectomy (CEA) operations to the prediction of neurological problems detected in the postoperative period. | 4 months
  Optic nerve sheath diameter measurement with USG is made using a high-frequency linear probe after the system settings are made suitable for the lens retina and vitreous body. It is performed by applying gel to the upper eyelid and placing the transducer in the temporal part of the eye, with the patient in a supine position with the head and body elevated 20-30 degrees.Optic nerve sheath diameter measurement with USG is made using a high-frequency linear probe after the system settings are made suitable for the lens retina and vitreous body. It is performed by applying gel to the upper eyelid and placing the transducer in the temporal part of the eye, with the patient in a supine position with the head and body elevated 20-30 degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- BasaksehirCamveSakuraSehirH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No